CLINICAL TRIAL: NCT07067697
Title: The Effect of Physical Exercise on the Physical Function of Hospitalized Older Adults Malnourished or at Risk of Malnourishment With Oral Nutritional Supplementation
Brief Title: Impact of Physical Exercise on Hospitalized Older Adults Malnourished or at Risk, With Oral Nutritional Support
Acronym: NUTPHYS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Miguel Servet (Other)
Collaborators: Nestle Health Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NUTPHYS
Record Dates: First submitted 2025-06-09; First posted 2025-07-16 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Hospitalized; Older Adults; Physical Exercise; Oral Nutritional Supplementation
Keywords: hospital-acquired disability; older adults; physical exercise; oral nutritional supplementation
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants included in this group will perform physical exercise
  Interventions: Other: Physical exercise
- Control (Active Comparator): Participants in this group will receive attention from a physiotherapist if needed.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Physical exercise — Progressive, supervised multicomponent physical exercise program, including aerobic resistance, strength, and balance training. Strength training for lower limbs (leg press and knee extension) and upper limbs (seated chest press) will be adapted to each individual's functional capacity.
  Arms: Intervention
Other: Usual Care — * Hospital physiotherapy for preventing nosocomial disability when necessary.
  * Hospital diet modifications appropriate to each participant's clinical situation.
  * Oral nutritional supplementation aimed at meeting daily nutritional requirements: 30 kcal/kg body weight, 1.5-2 g protein/kg body weight, 25 g daily fiber.
  * Approximate free water intake: women 1.5 L/day, men 2 L/day (unless clinically restricted).
  Arms: Control

SUMMARY:
The aim of this research is to analyze whether nutritional intervention combined with a multicomponent physical training program based on strength, balance, and aerobic exercises can prevent disability caused during hospitalization in individuals aged 75 years or older admitted for medical conditions, thereby improving functional and cognitive capacity.

To achieve this objective, we will conduct a randomized clinical trial in which patients are randomly assigned to either the control group, which does not perform the physical training, or the intervention group, which participates in the multicomponent physical training program.

DETAILED DESCRIPTION:
The main objective of the present study is to evaluate the differences in the impact of an intervention based solely on physical exercise on the functionality of hospitalized older patients, in an Acute Geriatric Unit, who are malnourished or at risk of malnutrition.

As secondary objectives:

1. To assess and compare changes in body composition following the intervention during hospitalization.
2. To evaluate and compare dietary intake, appetite progression, and food consumption throughout the intervention period.
3. To compare in-hospital infectious complications between the two groups.
4. To describe and compare changes in nutritional biochemical parameters between groups after the intervention and 30 days post-discharge.
5. To study changes in other physical function measures throughout the study period and compare them.
6. To describe the presence of molecular markers related to senescence and sarcopenia in patients and compare them between groups at discharge.
7. To study and compare changes in participants' cognitive status.
8. To evaluate and compare changes in perceived quality of life.
9. To assess and compare changes in maximal dynamic strength before and after the intervention.
10. To describe and compare hospital stays and 30-day readmission rates of study participants.
11. To describe participants' personal satisfaction with the intervention.
12. To describe the presence of potential side effects attributed to the intervention during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Aged 75 years or above
* Hospitalized in the Acute Unit of the Geriatrics Service at the University Hospital of Navarra
* 4 days or more of expected hospitalization
* Malnourished according to the GLIM criteria or at risk of malnourishment (MUST scale)
* Barthel Index ≥ 60 points
* Capable of tolerating oral intake
* Able to walk (with or without assistance)
* Able to understand instructions and communicate
* Consent to participate in the study after being informed of its objectives and who sign the informed consent (the participant or their legal guardian in case of disability).

Exclusion Criteria:

* Advanced major neurocognitive disorder (GDS 6 and 7)
* Uncontrolled cardiac arrhythmia, acute pulmonary thromboembolism, acute myocardial infarction, or bone fractures within the last 3 months
* Chronic kidney disease stage 4 or 5
* Safe and effective swallowing only with pudding texture
* Inability to participate in the physical exercise program due to physical limitations
* Participate in another study that may interfere with data interpretation or have participated in another study in six months prior to their entry into the study.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Function | Through study completion, an average of 4 days
  SPPB - Short Physical Performance Battery

SECONDARY OUTCOMES:
Anthropometrical Measurements | Through study completion, an average of 4 days
  Bioimpedance: PHASE ANGLE (PhA), Fat-Free Mass (FFM) and Muscle Mass (MM). Conventional and vectorial bioelectrical impedance analysis with a single-frequency bioelectrical impedance analyzer at 50 kHz (BIA 101 RJL, Akern Bioresearch, Florence, Italy)
Dietary intake | Through study completion, an average of 4 days
  Semi-quantitative questionnaire and a daily appetite assessment
Number and type of infectious complications | Through study completion, an average of 4 days
Nutritional status biomarkers | Through study completion, an average of 4 days, and 30 days post-discharge
  In blood: proteins, prealbumin, albumin, transferrin, lymphocytes, 25-hydroxyvitamin D, C-reactive protein.
Functional status | Through study completion, an average of 4 days, and 30 days post-discharge
  Barthel Index, Lawton Index
Frailty status | Baseline
  Linda Fried's Frailty Scale, from 0 to 5 (0 robust; 1,2 pre-frail; 3 to 5 frail).
Strength of upper and lower limbs | Through study completion, an average of 4 days
  Leg press, chest press, knee extension, and handgrip strength
Cognitive status | Through study completion, an average of 4 days
  Mini-Mental State Examination, 4AT
Affective status | Through study completion, an average of 4 days
  Yesavage's 15-item Geriatric Depression Scale (GDS-15)
Quality of life of participants | Through study completion, an average of 4 days
  EuroQoL-5D-3L
Adverse effects possibly attributed to the intervention | Through study completion, an average of 4 days

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Navarra, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No